CLINICAL TRIAL: NCT00441909
Title: Phase I Study of the Safety and Persistence of 0.1% UC-781 Vaginal Gel in HIV-1 Seronegative Women
Brief Title: Phase I Study of Safety and Persistence of UC-781 Vaginal Microbicide
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: CONRAD (Other)
Responsible Party: Sharon L. Hillier, PhD, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: U19AI051661 (NIH); U19AI051661 (NIH)
Record Dates: First submitted 2007-02-27; First posted 2007-03-01 (Estimated); Last update posted 2009-03-05 (Estimated); Status verified 2009-03

CONDITIONS: HIV Infections
Keywords: Anti-Infective Agents, Local; Healthy Women; Microbicides; UC-781; Vaginal Gel; HIV Seronegativity
MeSH Terms: conditions — HIV Infections | interventions — UC-781

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (8):
- 1A (Experimental): Participants will receive a single application of UC-781 vaginal microbicide, which will be inserted for 8 hours
  Interventions: Drug: UC-781
- 1B (Placebo Comparator): Participants will receive a single application of UC-781 vaginal microbicide placebo, which will be inserted for 8 hours
  Interventions: Drug: UC-781 placebo
- 2A (Experimental): Participants will receive a single application of UC-781 vaginal microbicide, which will be inserted for 4 hours
  Interventions: Drug: UC-781
- 2B (Placebo Comparator): Participants will receive a single application of UC-781 vaginal microbicide placebo, which will be inserted for 4 hours
  Interventions: Drug: UC-781 placebo
- 3A (Experimental): Participants will receive a single application of UC-781 vaginal microbicide, which will be inserted for 2 hours
  Interventions: Drug: UC-781
- 3B (Placebo Comparator): Participants will receive a single application of UC-781 vaginal microbicide placebo, which will be inserted for 2 hours
  Interventions: Drug: UC-781 placebo
- 4A (Experimental): Participants will receive a single application of UC-781 vaginal microbicide, which will be inserted for 0 hours
  Interventions: Drug: UC-781
- 4B (Placebo Comparator): Participants will receive a single application of UC-781 vaginal microbicide placebo, which will be inserted for 0 hours
  Interventions: Drug: UC-781 placebo

INTERVENTIONS:
Drug: UC-781 — 0.1% UC-781 Vaginal Gel
  Arms: 1A; 2A; 3A; 4A
Drug: UC-781 placebo — Vaginal Gel Placebo
  Arms: 1B; 2B; 3B; 4B

SUMMARY:
Vaginal microbicides are compounds that may protect women from HIV and other sexually transmitted infections (STIs). This study will determine the safety of the microbicide UC-781 by comparing the effects of keeping the microbicide in the vagina for different lengths of time.

DETAILED DESCRIPTION:
Vaginal microbicides are compounds applied to the inside of the vagina that may protect women against vaginal transmission of HIV and other STIs. This study will evaluate the safety of the vaginal microbicide UC-781. Studies have shown UC-781 to be an effective inhibitor of HIV-1 reverse transcriptase. UC-781 has been tested in animal models and in Phase I and II studies in humans. The results of these studies indicated that cervical tissue was fully protected from different variants of HIV. The purpose of this study is to assess the incidence of epithelial disruption and inflammation in the cervix, vagina, and vulva of healthy HIV uninfected women after a single exposure to UC-781 vaginal gel. This study will compare the results of leaving the microbicide in the vagina for varying lengths of time.

The duration of this study is approximately 35 days. Participants in this study will be randomly assigned to one of eight groups, and all participants will receive a single exposure of UC-781 or placebo gel. There will be five total study visits, including the screening and study entry visits. Screening will occur approximately 10 days prior to the study entry visit. At study entry, a single application of microbicide or placebo gel will be inserted for 0, 2, 4,or 8 hours in the vagina. Length of exposure time will differ, depending on which group a participant has been randomly assigned to. Following vaginal exposure to the microbicide, the microbicide will be rinsed off. Vaginal secretions will be collected to test antiviral activity against HIV and assess the amount of microbicide remaining in the vagina. Visits 3 through 5 occur at approximately 24 to 48 hours, 6 to 8 days, and 25 to 35 days following study entry.

At all visits, participants will be asked to complete a questionnaire and undergo a pelvic exam, STI tests, and vital signs measurements. Blood and urine collection will occur at each visit. On selected visits, a colposcopy will be conducted and participants will be interviewed regarding product acceptability, in addition to other measures. Between selected visits, participants will be asked to maintain sexual abstinence or use condoms.

ELIGIBILITY:
Inclusion Criteria for Screening Visit:

* HIV uninfected
* General good health
* Normal Pap smear within 12 months prior to screen or obtained at screening visit
* Anatomy that lends itself easily to visualization of the cervix
* Sexual abstinence (including vaginal, oral, and rectal) from Visit 1 to the completion of Visit 4
* Agree to use condoms provided by the study between Visits 4 and 5
* Agree to abstain from the use of intravaginal products or vaginal penetration throughout the study
* Willing to use acceptable forms of contraception until the completion of study
* Willing to participate in all study-related assessments and follow all study-related procedures

Inclusion Criteria for Study Entry:

* Meet all inclusion criteria for the screening visit at Study Entry
* Willing to stay in the Magee-Womens Hospital Clinical Research Center (MWH CRC) for up to 9 hours after gel insertion

Exclusion Criteria for Screening Visit:

* Menopause (at least 12 months without menses in absence of long-acting progestin use)
* Hysterectomy
* Latex allergy
* Use of a diaphragm, NuvaRing, or spermicide for contraception
* Diagnosed urogenital infection or suspected infection 21 days prior to study screening. More information on this criterion can be found in the protocol.
* Menses or other vaginal bleeding anticipated in the 17 days postscreening
* Antibiotic or antifungal therapy (vaginal or systemic) 14 days prior to study screening
* Injected nontherapeutic drugs 12 months prior to study screening
* Systemic immunosuppressive drug use 60 days prior to study screening
* Participation in drug, spermicide, and/or microbicide study 30 days prior to study screening
* Any condition that, in the opinion of the investigator, would interfere with the study
* Intravaginal use of any device or product (except tampons) 7 days prior to study screening
* Surgical procedure involving the pelvis in the 90 days prior to enrollment (e.g., dilation and curettage or evacuation, cervical biopsy, cryosurgery,any other surgery involving pelvic organs or area)
* Abnormal pelvic exam finding that, in the opinion of the investigator would complicate interpretation of the colposcopy
* Pregnancy, or within 90 days of last pregnancy
* Breastfeeding

Exclusion Criteria for Study Entry:

* Meets any of the exclusion criteria of the screening visit
* Diagnosed or suspected reproductive tract infection or urinary tract infection. More information on this criterion can be found in the protocol.
* Menses or other vaginal bleeding anticipated in the 8 days following study entry
* Injected nontherapeutic drugs between study screening and study entry
* Certain abnormal laboratory values

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2006-04; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Local and systemic safety of a one-time dose of UC-781 0.1 % gel for vaginal use at different durations of exposure in HIV uninfected women | Throughout study

SECONDARY OUTCOMES:
Persistence of UC-781 0.1% gel following a single application | At 0, 2, 4, or 8 hours post application
Systemic absorption of UC-781 following a single application of 0.1% UC-781 gel | At 0, 2, 4, or 8 hours post application
In vitro anti-HIV activity of cervicovaginal lavage fluid | Throughout study
Product acceptability | Throughout study
Measurement of vaginal flora characteristics | Throughout study
Changes in vaginal flora characteristics after a timed, single exposure | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Sharon L. Hillier, PhD, Principal Investigator — University of Pittsburgh; Harold C. Wiesenfeld, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Magee-Womens Hospital of University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Davis CW, Doms RW. HIV transmission: closing all the doors. J Exp Med. 2004 Apr 19;199(8):1037-40. doi: 10.1084/jem.20040426. Epub 2004 Apr 12. No abstract available. PMID 15078894
- [Background] Joshi S, Solomon S, Mayer K, Mehendale S. Preparing for efficacy trials of vaginal microbicides in Indian women. Indian J Med Res. 2005 Apr;121(4):502-9. PMID 15817959
- [Background] Keller MJ, Tuyama A, Carlucci MJ, Herold BC. Topical microbicides for the prevention of genital herpes infection. J Antimicrob Chemother. 2005 Apr;55(4):420-3. doi: 10.1093/jac/dki056. Epub 2005 Mar 2. PMID 15743896
- [Background] Minnis AM, Padian NS. Effectiveness of female controlled barrier methods in preventing sexually transmitted infections and HIV: current evidence and future research directions. Sex Transm Infect. 2005 Jun;81(3):193-200. doi: 10.1136/sti.2003.007153. PMID 15923284
- [Background] Weber J, Desai K, Darbyshire J; Microbicides Development Programme. The development of vaginal microbicides for the prevention of HIV transmission. PLoS Med. 2005 May;2(5):e142. doi: 10.1371/journal.pmed.0020142. Epub 2005 May 31. PMID 15916473